CLINICAL TRIAL: NCT02774772
Title: The Use of Home-monitoring and mHealth Systems to Predict Asthma Control and the Occurrence of Asthma Exacerbations
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: University of Manchester (Other); Imperial College London (Other); Leiden University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 15/NW/0845
Record Dates: First submitted 2016-02-24; First posted 2016-05-17 (Estimated); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators will collect a range of physiological, behavioural and environmental data using current mHealth and home-monitoring systems, environmental databases and patient characteristics, to determine to what extent asthma control and the occurrence of asthma exacerbations can be predicted.

DETAILED DESCRIPTION:
This observational study occurs alongside participants' normal asthma care. Participants will be asked to attend their normal GP and hospital appointments, and to continue to take their medication as determined by their usual healthcare team.

In addition to their normal care, participants will attend an induction visit and complete a 12-month home-monitoring period with 2 phases:

* Phase 1: one-month period of daily monitoring of asthma
* Phase 2: eleven-month period of weekly monitoring of asthma. Patients will be invited for a further 2-week period of daily monitoring between 2-9 months of Phase 2. The purpose of the second phase of daily monitoring is to assess the influence of seasonality (different seasons) on the patient's asthma.

  0 xxxx 1 ------ 2 ------ 3 ------ 4 yy-- 5 ------ 6------ 7 ------ 8 ------ 9 ------ 10 ------ 11 ----- 12

Figure 1. Schematic of study design. 0 1 2.., months; xxxx, first series of 4 weeks daily monitoring; ------ 11 months weekly monitoring; yy--, example of second series of 2 weeks daily monitoring during month 5 (the timing of this 2 weekly phase will be randomised over month 2-9).

A variety of measurements will be made at an induction visit and over the 12-month home-monitoring period, as detailed below:

Induction visit

Demographics - Age (yr), gender, nationality, ethnicity, body mass (kg), height (cm), body mass index (BMI), comorbidities, medication, previous moderate and severe asthma exacerbations in preceding 12 months, previous severe asthma exacerbations requiring hospital attendance / admission (No in preceding 12 months), number of intensive care admission for asthma (ever), smoking history and social economic status.

Questionnaires

* Asthma control will be assessed by the Asthma Control Questionnaire (ACQ). [A patient's asthma control status will be classified as Controlled (ACQ≤0.75), Partly Controlled (0.75<ACQ≤1.5) or Uncontrolled (ACQ>1.5)].
* The typical diet of participants will be assessed via the Global Allergy and Asthma European Network (GA2LEN) food frequency questionnaire.
* Sinusitis/rhinoconjunctivitis will be determined via the Sino-Nasal Outcome Test 22 (SNOT 22)
* Anxiety and depression will be determined via the hospital anxiety and depression score (HADS)
* Characteristics such as health directed behaviours and self-monitoring will be determined using the Health education impact Questionnaire (HeiQ)
* Mini-Asthma Quality of Life Questionnaire (mini-AQLQ)

Clinical tests

- Atopic status will be determined via previous skin-prick test or blood test results.

(If a patient's atopic status is unknown, a standard skin-prick test or blood test will be conducted).

* The diagnosis of asthma will be verified via a previous test result, using one of the following; a bronchodilator reversibility test, one-week peak flow monitoring or a bronchial challenge test. (If a patient's asthma diagnosis has not been verified from one of the tests listed above, they may be performed at screening visits)
* Lung function (spirometry) will be conducted according to ERS guidelines
* Airways inflammation will be determined by the level of Fractional exhaled Nitric Oxide (FeNO) according to established guidelines
* Exhaled Breath Temperature, as measured by the X-halo device

Phase 1 (first 4-week daily monitoring)

The measurements in Phase 1 will be collected during the first 4 weeks of monitoring, and will be self-administered by the participant. Measurements will occur continuously, daily, weekly or less frequent, as specified below:

Questionnaires

* Daily, Asthma Control Diary (ACD)
* Daily, online medication diary
* Weekly, assessment of the occurrence of exacerbation, determined by a custom questionnaire.
* Monthly, mini Asthma Quality of Life Questionnaire (mini-AQLQ)
* Sinusitis will be determine via the SNOT 22 at the end of the first 4-week daily monitoring
* Technology acceptance via ASQ at the end of the first 4-week daily monitoring 25

Physiological monitoring

* Continuous data collection, via wearable sensors
* Pulse, exercise level via Fitbit HR wristband
* Medication usage and adherence via Smartinhaler device in a subset of 60 participants
* Measurement of breath rate via Spire device
* Daily, twice daily home spirometry (FEV1) via Piko-1 device
* Daily, twice-daily Fractional exhaled Nitric Oxide (FeNO) via NIOX-VERO device in a subset of 60 participants
* Daily, twice-daily Exhaled Breath Temperature (EBT) via X-halo device, in a subset of 60 participants

Environmental

* Retrospective collection of environmental conditions for patients home and work address, including:
* Ozone (O3)
* air pollution (PM10, PM2.5)
* ambient temperature
* Nitrous oxide (NO2)
* Sulphur dioxide (SO2)
* Weather conditions
* Mean temperature
* Humidity
* Pollen counts

Phase 2 (month 2-12) The measurements in Phase 2 will occur continuously, weekly or less frequent, as specified below. The weekly measurements will occur on a fixed day of the week, determined by participants for convenience, and all the measurements will be self-administered by the participant.

Questionnaires

* Weekly online Asthma Control Questionnaire
* Weekly assessment of the occurrence of exacerbation, determined by a custom questionnaire.
* Weekly, medication diary (custom made questionnaire)
* Monthly mini Asthma Quality of Life Questionnaire (mini AQLQ)
* Monthly, Sinus symptoms will be determine via the SNOT 22 questionnaire
* Technology acceptance via ASQ at 6 and 12 months
* Global Allergy and Asthma European Network (GA2LEN) food frequency questionnaire will be completed at the end of the study.

Physiological monitoring

* Continuous data collection, via wearable sensors
* Pulse, exercise level via Fitbit HR wristband
* Medication usage and adherence via Smartinhaler device in a subset of 60 participants
* Measurement of breath rate via Spire device
* Weekly, home spirometry (FEV1) via Piko-1
* Weekly, Fractional exhaled Nitric Oxide (FeNO) by NIOX-VERO in a subset of 60 participants
* Weekly, Exhaled Breath Temperature (EBT) by X-halo, in a subset of 60 participants

Environmental

- Retrospective collection of environmental conditions for patients home and work address, as detailed above.

A second series daily monitoring (as described in phase 1) will be performed over a two week period, randomised between 2 to 9 months.

ELIGIBILITY:
Inclusion Criteria:

1. Doctors-diagnosis of asthma with confirmation of asthma from one or more of the following tests in medical notes:

   i) Reversibility of 12% and 200ml in a spirometry following administration of a bronchodilator medication ii) Peak flow monitoring for one week iii) Positive bronchial challenge
2. BTS asthma treatment step 2-4, for a minimum of 6 months in the previous year
3. A course of oral prednisone for a minimum of three days, or an emergency department visit/hospitalisation for asthma, in the previous twelve months. Or currently experiencing uncontrolled asthma (based on the result of the Asthma Control Questionnaire)

Exclusion Criteria:

1. Comorbidities that cause overlapping symptoms such as breathlessness, wheeze, cough or other interfering chronic condition (for example other symptomatic chronic respiratory disease, cardiac failure etc.).
2. Unable to understand English or Dutch, as appropriate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One hundred and fifty patients with asthma will be recruited from outpatient clinics and from general practices in London, Manchester (United Kingdom) and Leiden (Netherlands).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Asthma control using the asthma control diary | After 1 month
  A score of 0.0-0.75 is classified as well-controlled asthma; 0.75-1.5 as a partly controlled; and >1.5 as poorly controlled asthma.
Severe asthma exacerbations | 1 year & preliminary analysis after 1 month
  Severe asthma exacerbations are events that require urgent action on the part of the patient and physician to prevent a serious outcome, such as hospitalization or death from asthma. The occurrence of severe asthma exacerbations is an important marker of poor asthma control. Severe asthma exacerbations are defined by the occurrence of at least one of the following:
  * Use of systemic corticosteroids (tablets, suspension, or injection), or an increase from a stable maintenance dose, for at least 3 days. For consistency, courses of corticosteroids separated by 1 week or more should be treated as separate severe exacerbations.
  * A hospitalisation or ER visit because of asthma, requiring systemic corticosteroids.
Moderate asthma exacerbations | 1 year & preliminary analysis after 1 month
  A moderate asthma exacerbation is an event that, when recognized, should result in a temporary change in treatment, in an effort to prevent the exacerbation from becoming severe. Moderate asthma exacerbations are defined by occurrence of at least one or more of the following:
  * deterioration in symptoms,
  * deterioration in lung function,
  * and increased rescue bronchodilator use. These features should last for 2 days or more, but not be severe enough to warrant systemic corticosteroid use and/or hospitalization. ER visits for asthma (e.g., for routine sick care), not requiring systemic corticosteroids, are also classified as moderate exacerbations

SECONDARY OUTCOMES:
User acceptence | 1 year & preliminary analysis after 1 month
  User acceptance of each mHealth and home-monitoring system, as determined by user-adherence and the After-Scenario Questionnaire feedback (ASQ)
Asthma Control using asthma control questionnaire | 1 year
  A score of 0.0-0.75 is classified as well-controlled asthma; 0.75-1.5 as a partly controlled; and >1.5 as poorly controlled asthma.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of South Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Khusial RJ, Sont JK, Usmani OS, Bonini M, Chung KF, Fowler SJ, Honkoop PJ. The Effect of Inhaled Beta-2 Agonists on Heart Rate in Patients With Asthma: Sensor-Based Observational Study. JMIR Cardio. 2024 Dec 11;8:e56848. doi: 10.2196/56848. PMID 39661964
- [Derived] Honkoop PJ, Simpson A, Bonini M, Snoeck-Stroband JB, Meah S, Fan Chung K, Usmani OS, Fowler S, Sont JK. MyAirCoach: the use of home-monitoring and mHealth systems to predict deterioration in asthma control and the occurrence of asthma exacerbations; study protocol of an observational study. BMJ Open. 2017 Jan 24;7(1):e013935. doi: 10.1136/bmjopen-2016-013935. PMID 28119390